Data analysis will adhere closely to the Consolidated Standards of Reporting Trials guidelines. Analysis will follow the intention-to-treat principle in which subjects will be analyzed in the group to which they were randomized, regardless of whether or not they received the assigned intervention. This is important because analysis according to the intention-to- treat principle is accepted as the most unbiased assessment of the true therapeutic benefits of a treatment. A per protocol Analysis will be performed as well. There are no planned interim analyses.

We will first compare baseline characteristics and demographics of the two groups at. Formal statistical testing will be limited to selected baseline characteristics considered to be prognostic factors for the primary outcome such as mode of delivery, antepartum blood pressures, and presence or absence of chronic hypertension. The Chi-squared or Fisher's exact tests will be used as appropriate to compare the primary outcome (proportion of subjects requiring antihypertensive medications at discharge) and other categorical secondary outcomes and prognostic factors between trial groups. Relative risks and confidence intervals associated with the primary and categorical secondary outcomes will be calculated and reported. Distribution of continuous prognostic factors and secondary outcome measures will be assessed by visual inspection of histograms and the Kolmogorov-smirnov test. Normally distributed variables will be compared by using the two-group independent t-test. If variables are not normally distributed, the Mann-Whitney U test will be used to make comparisons between the trial groups

A stepwise logistic regression model will be used to identify and estimate the effect of multiple prognostic factors on the probability of need for antihypertensive at time of discharge and other categorical outcomes.

Additional interaction analyses, using the Brewlow-Day test, for the primary outcome will be performed for the following subgroups:

- 1) Presence of chronic medical conditions
  - a. Patients with hypertensive disorders prior to pregnancy
  - b. Patients with diabetes mellitus (gestational diabetes, T1DM, T2DM)
- 2) Patients with mild renal dysfunction (Cr >1.1 and CrCl >60 mL/min)
- 3) Patients with prolonged antepartum diagnosis of preeclampsia
- 4) Patients requiring scheduled antihypertensive medications prior to delivery
- 5) Gestational age at delivery
- 6) Race
- 7) BMI